CLINICAL TRIAL: NCT04896554
Title: Comparison of the Health Literacy of Our Patients Who Quit Smoking and Who Cannot Quit Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Seyhan Dülger,MD, associate professor, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011-KAEK-25 2021/05-01
Record Dates: First submitted 2021-05-07; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Smoking Cessation; Health Literacy
Keywords: smoking cessation; health literacy
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- quit smoking (Active Comparator): patients who have quit smoking
  Interventions: Behavioral: Health literacy scale
- not quit smoking (Active Comparator): patients who have not quit smoking
  Interventions: Behavioral: Health literacy scale

INTERVENTIONS:
Behavioral: Health literacy scale — The Turkish version of The European Health Literacy Survey (HLS-EU) Health Literacy Questionnaire scale (ASOY-TR) was used to measure health literacy. This scale consists of 47 questions. Each item has 4 degrees such that 1 = Very difficult, 2 = Difficult, 3 = Easy, 4 = Very easy. Code 5 is used for the expression "I don't know". The total score that can be obtained from the scale is between 47-188. For the sake of ease of calculation, the total score is standardized with the following formula to take a value between 0-50.
  Formula = Index = (arithmetic mean-1) x [50/3] High score means better health literacy.

SUMMARY:
The aim of the study was determined to examine the relationship between the health literacy scales of the patients who came to the smoking cessation clinic and their smoking cessation success.

The patient follow-up files registered in the archive of the smoking cessation clinic will be scanned for the last 2 years and the demographic data and follow-up information of the patients will be reached. Patients who have completed the 1-year follow-up period will be contacted by phone, questioning whether they smoke or not, and will be invited to answer the health literacy scale. Accepting patients will be divided into two groups as those who quit smoking and those who cannot, and health literacy scales will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who applied to the smoking cessation clinic for smoking cessation
2. over the age of 18
3. Those who agree to answer the health literacy scale form

Exclusion Criteria:

1. Patients under the age of 18
2. Those who do not agree to answer the health literacy scale form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Health literacy | After 1 year of follow-up in the smoking cessation clinic
  The Turkish version of The European Health Literacy Survey (HLS-EU) Health Literacy Questionnaire scale (ASOY-TR) was used to measure health literacy. This scale consists of 47 questions. Each item has 4 degrees such that 1 = Very difficult, 2 = Difficult, 3 = Easy, 4 = Very easy. Code 5 is used for the expression "I don't know". The total score that can be obtained from the scale is between 47-188. For the sake of ease of calculation, the total score is standardized with the following formula to take a value between 0-50.
  Formula = Index = (arithmetic mean-1) x [50/3] High score means better health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Seyhan Dülger, Principal Investigator — Bursa Yüksek İhtisas Education And Training Hospital
Locations (1):
- Bursa Yüksek İhtisas EAH, Bursa, Eyalet/Yerleşke, Turkey (Türkiye)